CLINICAL TRIAL: NCT07236359
Title: A Randomised Control Trial Evaluating Well Being and Patient Reported Outcomes After Robotic Single-port Nipple Sparing Mastectomy and Implant Reconstruction
Brief Title: Evaluation of Well Being and Patient Reported Outcomes After Robotic Single-port Nipple Sparing Mastectomy and Implant Reconstruction
Acronym: Reborn-i
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Arnold Hill, Professor, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25/72
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Reconstruction; Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2); Robotic Surgery
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port robotic nipple-sparing mastectomy with immediately implant based reconstruction. (Experimental): Intervention
  Interventions: Procedure: Intervention
- Standard open nipple sparing mastectomy with immediate implant-based reconstruction. (Active Comparator): Standard of care
  Interventions: Procedure: Standard open nipple sparing mastectomy with immediate implant-based reconstruction

INTERVENTIONS:
Procedure: Intervention — Single-port robotic nipple-sparing mastectomy with immediately implant based reconstruction.
  Arms: Single-port robotic nipple-sparing mastectomy with immediately implant based reconstruction.
Procedure: Standard open nipple sparing mastectomy with immediate implant-based reconstruction — Standard open nipple sparing mastectomy with immediate implant-based reconstruction
  Arms: Standard open nipple sparing mastectomy with immediate implant-based reconstruction.

SUMMARY:
This study is being carried out to better understand how different types of mastectomy surgeries affect women's recovery, satisfaction, and overall well-being after breast cancer surgery and reconstruction. There are different ways to perform a mastectomy. In some patients, a nipple-sparing mastectomy may be suitable, where the nipple and surrounding breast skin are preserved. This approach allows for immediate breast reconstruction with an implant, which is placed at the same time as the mastectomy to restore the breast shape. A newer technique called robotic single-port nipple-sparing mastectomy uses advanced robotic technology to remove breast tissue through a small hidden incision at the side of the chest. This method may reduce scarring, pain, and recovery time, while preserving the appearance and sensation of the breast.

However, while early studies suggest this technique is safe and effective, more evidence is needed to compare it directly with standard surgeries.

This study will compare:

* Robotic nipple-sparing mastectomy
* Standard (open) nipple-sparing mastectomy We will assess patient satisfaction, body image, physical and emotional well-being, and surgical outcomes over 12 months following surgery. By taking part, you are helping researchers evaluate whether robotic and nipple-sparing approaches offer measurable benefits to patients.

Taking part in this study will not affect your surgery or the care you receive. You will be given the best treatment available based on your individual medical needs, whether or not you decide to participate in the research.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Candidates who have already been selected to undergo nipple sparing mastectomy and immediate implant reconstruction by the breast MDT for the following indications:
* Genetic mutation carriers undergoing risk-reducing mastectomy.
* Ductal carcinoma in situ (DCIS) requiring mastectomy.
* Early invasive breast cancer requiring mastectomy.
* The tumour must not have skin involvement and no evidence of invasive disease within 1cm of skin, nipple or Pec major muscle (as proven on MRI).
* Candidates for immediate breast reconstruction with IMPLANT reconstruction
* Fluent in English
* Fit for general anaesthetic
* Signed informed consent form

Exclusion Criteria:

* Advanced breast cancer with skin involvement.
* Nipple involvement for Nipple Sparing Mastectomy Arms.
* Prior chest wall radiation therapy
* Pregnancy
* Lactation
* Patients with insufficient English to sign an informed consent (i.e. interpreter required).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Secondary Outcome Measures | 1 year
  * Surgical complication rates within 30 and 90 days, classified according to the Clavien-Dindo system.
  * Reoperation rates and need for unplanned return to theatre.
  * Length of hospital stay and drain duration
  * Operative time and estimated intraoperative blood loss.
  * Time to return to daily activities including work and physical exercise.
  * Aesthetic outcomes, assessed both by patient-reported satisfaction and by an independent panel review of standardized postoperative photographs.
  * Oncologic outcomes, including final pathology margin status and local recurrence (if applicable during follow-up).
  * Amount of residual breast tissue left on post operative MRI at 6 months in the different groups.
Primary Outcome Measure | 1 year
  The primary endpoint of this study is the difference Breast Q scores at 12 months.

IPD SHARING:
Plan to Share IPD: Yes
Protocol and anonymous study data will be shared through peer reviewed publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Toesca A, Sangalli C, Maisonneuve P, Massari G, Girardi A, Baker JL, Lissidini G, Invento A, Farante G, Corso G, Rietjens M, Peradze N, Gottardi A, Magnoni F, Bottiglieri L, Lazzeroni M, Montagna E, Labo P, Orecchia R, Galimberti V, Intra M, Sacchini V, Veronesi P. A Randomized Trial of Robotic Mastectomy Versus Open Surgery in Women With Breast Cancer or BrCA Mutation. Ann Surg. 2022 Jul 1;276(1):11-19. doi: 10.1097/SLA.0000000000004969. Epub 2021 Jun 9. PMID 34597010
- [Background] Sarfati B, Honart JF, Leymarie N, Rimareix F, Al Khashnam H, Kolb F. Robotic da Vinci Xi-assisted nipple-sparing mastectomy: First clinical report. Breast J. 2018 May;24(3):373-376. doi: 10.1111/tbj.12937. Epub 2017 Dec 18. PMID 29251382